CLINICAL TRIAL: NCT00622583
Title: A Two-Year Follow-up, Post-Implantation, Multi-center, International Hernia Mesh Registry
Brief Title: International Hernia Mesh Registry
Acronym: IHMR
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-06-007
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Hernia
Keywords: Herniorrhaphy
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation Group: Subjects who meet the inclusion/exclusion criteria who have had a hernia repair.

SUMMARY:
This is an open-label, multi-center, long-term, prospective hernia mesh registry. A minimum of 4,800 hernia patients will be enrolled from approximately 60 active sites globally

DETAILED DESCRIPTION:
Patients will be followed for 2-years post-implantation, in a post-market setting to help identify best practices leading to lower recurrence rates and decreases in chronic pain, associated with the hernia repair procedure.

ELIGIBILITY:
Inclusion Criteria

Patients must satisfy the following criteria before entering the registry:

1. Provide written informed consent prior to surgery;
2. Male or female patients that are > 18 years of age;
3. Be literate and able to understand a language available in the Registry Patient Questionnaires;
4. Scheduled to receive a surgically implanted ETHICON synthetic mesh using any fixation method or a non-ETHICON synthetic mesh which must be fixated with SECURESTRAP® or SECURESTRAP® Open for repair of a hernia defect;
5. Agree to provide long-term, outcomes data to Quintiles Outcome;
6. Agree to provide contact information;
7. Two or more pieces of the same mesh product sewn together will be considered as one mesh, and is therefore allowed in this registry

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from participating in the registry:

1. Patients that are <18 years of age;
2. Patients who have been entered into the registry previously;
3. Employees of the investigator or registry center with direct involvement in the proposed registry or other studies under the direction of that investigator or registry center and employees of ETHICON;
4. Patients suffering from and currently receiving medication for chronic pain (defined as suffering pain for greater than 3 months);
5. Patients known to be suffering from pre-existing chronic depression;
6. Patients currently known or suspected to abuse drugs or alcohol;
7. Patients suffering from a terminal illness (e.g. cancer);
8. Patients requiring multiple hernia repairs (including bilateral inguinal/femoral);
9. Patients requiring any other (concomitant) surgical procedure;
10. Patients suffering from an ongoing infection, sepsis, contaminated mesh or fistulas;
11. Patients who require hiatal, paraesophageal or diaphragmatic hernia repair;
12. Patients requiring two different types of meshes;
13. Patients requiring two or more meshes not sewn together
14. Patients scheduled to receive a surgically implanted biologic mesh product for repair of a hernia defect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic and patients of the investigators at local clinics or hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 5179 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Recurrence of the hernia | 1 month, 6-months, 12 months, 2 years
Pain assessment scores by patients for the duration of the registry (Acute pain and Chronic pain) | 1 month, 6-months, 12 months, 2 years

SECONDARY OUTCOMES:
Assessment of post-operative complications/safety | At the time of surgery
Assessment of procedure time | At the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Niels-Derrek Schmitz, M.D., Study Director — Ethicon, Inc.
Locations (54):
- United States (18):
  - Florida Hospital Celebration Health, Celebration, Florida
  - Center for Hernia Repair, Sarasota, Florida
  - Steward Norwood Hospital, Norwood, Massachusetts
  - University of Missouri-Columbia, Columbia, Missouri
  - SurgiCare of Missouri, P.C., Jefferson City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Queens Long Island Medical Group, Hicksville, New York
  - Laparoscopic Surgical Center of New York, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Owen Drive Surgical Clinic of Fayetteville, Fayetteville, North Carolina
  - Pinehurst Surgical Center, Pinehurst, North Carolina
  - South East Area Health Education Center (SEAHEC), Wilmington, North Carolina
  - Southwest Specialty Clinics, Oklahoma City, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - North Penn Surgical Associates, Lansdale, Pennsylvania
  - Dallas Hernia Institute, Duncanville, Texas
  - Kirby Surgical Center, Houston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
- Australia (3):
  - Queen Elizabeth Hospital, Woodville, South Australia
  - MercyCare Mount Lawley Hospital, Mount Lawley, Western Australia
  - The Wesley Hospital, Auchenflower
- Belgium (2):
  - Imelda Hospital, Bonheiden
  - University Hospital Ghent, Ghent
- Canada (3):
  - Centre for the Advancement of Minimally Invasive Surgery (CAMIS), Edmonton, Alberta
  - Hamilton Health Sciences - General, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
- Huadong Hospital- Affilated to Fudan University, Shanghai, China
- France (10):
  - Hopital Prive D'Antony, Antony
  - CH Avignon - Service de Chirurgie Digestive, Avignon
  - CHU Hotel Dieu, Clermont-Ferrand
  - Hospital Saint Philibert, Lomme
  - Hopital Prive Mermoz, Lyon
  - HIA Laveran, Marseille
  - CHU de Nancy, Nancy
  - Service de Chirurgie Generale et Cancerologie Digestiv, Nice
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Centre Hospitalier Robert Debre, Reims
- Lukaskrankenhaus, Neuss, Germany
- Universita Cattolica Sacro Cuore, Rome, Italy
- Jeroen Bosch Hospital, 's-Hertogenbosch, Netherlands
- New Somerset Hospital, Cape Town, South Africa
- Spain (2):
  - San Augustin De Aviles Hospital, Avilés
  - University Hospital Virgen del Rocio, Seville
- Sodertalje Hospital, Södertälje, Sweden
- United Kingdom (10):
  - Hinchingbrooke Hospital, Huntingdon, Cambrideshire
  - Royal United Hospital, Bath, Somerset
  - University Hospitals of North Midlands, Stoke-on-Trent, Staffordshire
  - Ayr Hospital, Ayr
  - Dorset County Hospital, Dorchester
  - Royal Bolton Hospital, Farnworth
  - St Mary's Hospital, London
  - North Tyneside General Hospital, North Shields
  - Northampton General Hospital, Northampton
  - Royal Alexandra Hospital, Paisley